CLINICAL TRIAL: NCT00613522
Title: Role of Nocturnal Respiratory Disorders on Ischemic Stroke Occurrence
Brief Title: Role of Obstructive Sleep Apnea in Stroke Appearance
Acronym: AVSAS
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX2006/10; 2007-A00382-51
Record Dates: First submitted 2008-01-30; First posted 2008-02-13 (Estimated); Last update posted 2015-03-05 (Estimated); Status verified 2015-03

CONDITIONS: Stroke; Obstructive Sleep Apnea
Keywords: Sleep apnea, Berlin, Stroke
MeSH Terms: conditions — Stroke; Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- case: Fist ischaemic hemispheric stroke or TIA
  Interventions: Other: polygraphic study
- control: No ischaemic hemispheric stroke or TIA
  Interventions: Other: polygraphic study

INTERVENTIONS:
Other: polygraphic study — Berlin scale will be measured. A polygraphic study will be performed to subjects with a Berlin scale > 2.
  Patients stroke characteristics will be recorded (initial severity, stroke mechanism) at baseline and stroke outcome will be evaluated at 3 months (stroke recurrence and functional outcome).
  Controls will be evaluated at 3 months using a phone interview

SUMMARY:
Stroke is the third leading cause of death in industrialized countries and the first cause of handicap in adults. Several stroke risk factors were identified such as high blood pressure, diabetes mellitus, hypercholesterolemia or cardiac arrhythmias. Sleep respiratory disorders have been found to be frequent among patients with stroke. Among them obstructive sleep apnea (OSA) syndrome seems to be the most important due to its association with high blood pressure and atrial fibrillation.

Stroke can be responsible of central apneas, therefore the differential diagnosis between central apneas and pure OSA after stroke is sometimes difficult. The misidentification of OSA can explain the poor tolerance of CPAP treatment by these patients. The purpose of the present study is to investigate the association between pre-stroke OSA syndrome OSA diagnosed on specific scales and confirmed by polygraphic studies and stroke occurrence.

DETAILED DESCRIPTION:
• Principal Objective : Investigate the association between obstructive sleep apnea diagnosed and hemispheric ischemic stroke

• Secondary Objective :

Evaluate the relation between obstructive sleep apnea and:

* stroke mechanisms
* stroke prognosis
* post-stroke tolerance to CPAP treatment.

  * Study design :

Prospective case-control study

• Inclusion criteria :

Patients (150):

Fist ischaemic hemispheric stroke or TIA Age: 50 to 90 French native speaker Able to answer the questions

Controls (600):

Age: 50 to 90 French native speaker Able to answer the questions

• Exclusion criteria : Patients Haemorrhagic stroke Stroke of the brainstem Past medical history of ischaemic stroke Dementia Confusion Unable to give his informed consent

Controls:

Past medical history of ischaemic stroke Dementia Confusion Unable to give his informed consent

• Study plan: Cases will be recruited in the stroke unit of the Pr Orgogozo at the Bordeaux University hospital. After verification of inclusion and exclusion criteria Berlin scale will be measured. A polygraphic study will be performed to patients with a Berlin scale > 2. Patients stroke characteristics will be recorded (initial severity, stroke mechanism) at baseline and stroke outcome will be evaluated at 3 months (stroke recurrence and functional outcome).

Controls will be recruited among sex and age matched patients hospitalized at the Bordeaux-University hospital for investigation of non-vascular disorder. After verification of inclusion and exclusion criteria Berlin scale will be measured. A polygraphic study will be performed to subjects with a Berlin scale > 2. Controls will be evaluated at 3 months using a phone interview

• Number of subjects : 150 cases and 600 controls

ELIGIBILITY:
Inclusion criteria (patients) :

* Fist ischaemic hemispheric stroke or TIA
* Age: 50 to 90
* French native speaker
* Able to answer the questions

Inclusion criteria (Controls):

* Age: 50 to 90
* French native speaker
* Able to answer the questions

Exclusion criteria (patients):

* Haemorrhagic stroke
* Stroke of the brainstem
* Past medical history of ischaemic stroke
* Dementia
* Confusion
* Unable to give his informed consent

Exclusion criteria (Controls):

* Past medical history of ischaemic stroke
* Dementia
* Confusion
* Unable to give his informed consent

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cases will be recruited in the stroke unit at the Bordeaux University hospital Controls will be recruited among sex and age matched patients hospitalized at the Bordeaux-University hospital for investigation of non-vascular disorder
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2007-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Stroke recurrence | 3 months

SECONDARY OUTCOMES:
Stroke outcome (Rankin, Barthel) Stroke mechanism CPAP tolerance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc ORGOGOZO, MD, Principal Investigator — University Hospital, Bordeaux
Locations (1):
- Groupe Hospitalier Pellegrin - Place Amélie Raba Léon, Bordeaux, France